CLINICAL TRIAL: NCT06526000
Title: Retrospective EMR Study to Assess Changes in Immunoglobulins in Patients With Relapsing Forms of Multiple Sclerosis Treated With Anti-CD20 Monoclonal Antibodies
Brief Title: Study to Assess Changes in Immunoglobulins in Patients With Relapsing Multiple Sclerosis Treated With Anti-CD20 Therapies
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: COMB157GUS26
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Relapsing Multiple Sclerosis; Clinically Isolated Syndrome; Relapsing-remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Relapsing Multiple Sclerosis Cohort: Patients with relapsing forms of multiple sclerosis who had newly initiated anti-CD20 treatment after March 2017.

SUMMARY:
This was an observational retrospective cohort study using electronic medical records (EMRs) to study immunoglobulin levels over time among patients with relapsing forms of multiple sclerosis (MS) newly initiating anti-CD20 monoclonal antibody treatment in clinical practice.

The index date was defined as the date of anti-CD20 drug initiation during the study period. The baseline period was defined as 12 months prior to the index date.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 years or older at index.
* Patients with RMS, including clinically isolated syndrome (CIS), relapsing-remitting multiple sclerosis (RRMS), and secondary progressive multiple sclerosis (SPMS) at the time of initiating anti-CD20 treatment.
* Newly initiated anti-CD20 treatment after March 2017 (no history of anti-CD20 therapy at any time in medical record before this date) to the latest data cutoff (November 2022).
* Patients with at least one documented IgG lab value pre- and post-anti-CD20 drug initiation.

Exclusion criteria:

* Patients with diagnosis of primary progressive multiple sclerosis (PPMS) prior to anti-CD20 treatment.
* Participated in an anti-CD20 drug clinical trial during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage Change per Year in Immunoglobulin G (IgG) Levels in Patients Receiving Ocrelizumab | Up to 5 years

SECONDARY OUTCOMES:
Percentage of Patients Newly Treated with Ocrelizumab With Low Immunoglobulin Values | Up to 5 years
  Low immunoglobulin values were defined as greater than or equal to 1 immunoglobulin G (IgG) lab value of less than 500 milligrams per deciliter (mg/dL) or greater than or equal to 1 immunoglobulin M (IgM) lab value of less than 25 mg/dL.
Percentage Change per Year in Immunoglobulin M (IgM) Levels in Patients Receiving Ocrelizumab | Up to 5 years
Percentage Change per Year in IgG Levels Associated With Risk Factors in Patients Treated With Ocrelizumab | Up to 5 years
  Risk factors included: age and disease duration.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States